CLINICAL TRIAL: NCT07108907
Title: ORANGE- TEER (Outcome Registry and Assessment of New Edge-to-Edge Repair)
Brief Title: Outcome Registry and Assessment of New Edge-to-Edge Repair
Acronym: ORANGE-TEER
Status: Recruiting | Type: Observational
Sponsor: Abby Geerlings (Other)
Responsible Party: Sponsor-Investigator, Abby Geerlings, PhD Candidate, MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: 2025.0301
Record Dates: First submitted 2025-07-25; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Mitral Regurgitation
Keywords: Mitraclip
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mitraclip: all patients receiving a mitraclip

SUMMARY:
The goal of this observational study is to learn about the long-term effects of Edge-tot-edge repair of all the patients of AmsterdamUMC, to treat their Mitral regurgitation (MR). The main question it aims to answer is:

The patient selection process could be optimized. Participants are already receiving edge-to-edge repair as part of their standard medical care and will additionally complete quality-of-life survey questions.

DETAILED DESCRIPTION:
Mitral regurgitation (MR) affects more than 10% of individuals over the age of 75, and with an aging population, its prevalence is expected to continue rising in the coming years. Treatment options include surgical repair, surgical replacement, medical therapy, cardiac resynchronization therapy (CRT), or transcatheter valve repair. For percutaneous mitral valve repair, the transcatheter edge-to-edge repair (M-TEER) technique is the preferred approach. This technique involves the use of the MitraClip (Abbott) and PASCAL (Edwards) devices, which are derived from the surgical Alfieri technique.

Since 2009, the M-TEER procedure has been performed in patients who, based on assessment by the heart team and mitral valve team, are deemed unsuitable for surgery but are eligible for this percutaneous treatment.

Using data from all patients undergoing M-TEER at Amsterdam UMC, the investigators aim to conduct research focused on improving patient selection and alleviating symptoms associated with mitral valve disease.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

* Age ≥ 18 years
* Accepted for M-TEER (Minimally Invasive Transcatheter Edge-to-Edge Repair) procedure

Exclusion Criteria:

- Unable to complete the questionnaires

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients recieving a M-TEER procedure
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline and 6 months
  Change in health-related quality of life as assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline to 6 months. The KCCQ is a validated, disease-specific instrument measuring physical function, symptoms, social limitations, and quality of life in patients with heart failure. Scores range from 0 to 100, with higher scores indicating better health status.
  Unit of Measure: KCCQ score (0-100)
Change in quality of life measured by the 36-Item Short Form Survey (SF-36) | Baseline and 6 months
  Change in health-related quality of life as assessed by the 36-Item Short Form Survey (SF-36) from baseline to 6 months. The SF-36 is a validated, generic instrument assessing physical and mental health across 8 domains. Scores are standardized to a 0-100 scale, with higher scores indicating better perceived health.
  Unit of Measure: SF-36 score (0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No